CLINICAL TRIAL: NCT05280015
Title: A Phase II, Prospective, Multicenter Study Assessing the Contribution and Tolerance of a Multi-targeted Microbiotherapy in Addition to Venlafaxine, After Failure of a First-line Antidepressant Treatment in Depressed Patients
Brief Title: Microbiotherapy in Characterized Depressive Disorder
Acronym: PROMOOD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Fondation FondaMental (Other); GYNOV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021/621
Record Dates: First submitted 2022-02-18; First posted 2022-03-15 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Depression; Depressive Disorder; Depressive Disorder, Major
Keywords: depression; microbiotherapy
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: After randomization, subjects suffering of MDD and treated by venlafaxine in a second-line assigned to start the microbiotherapy pr placebo during 12 weeks. The microbiotherapy is GynMDD developped by Gynov and which is composed by a probiotic associated to polyphenol and an amino acid.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbiotherapy in addition of venlafaxin (Active Comparator): Subjects suffering of MDD and treated by venlafaxine in a second-line assigned to start the microbiotherapy during 12 weeks. The microbiotherapy is GynMDD devlopped by Gynov and which is composed by a probiotic associated to polyphenol and an amino acid.
  Interventions: Dietary Supplement: microbiotherapy (GynMDD)
- calibration arm (Placebo Comparator): Subjects suffering of MDD and treated by venlafaxine in a second-line assigned to start the placebo therapy during 12 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: microbiotherapy (GynMDD) — multi-target microbiotherapy add-on venlafaxine
  Arms: Microbiotherapy in addition of venlafaxin
Other: placebo — placebo add-on venlafaxine
  Arms: calibration arm

SUMMARY:
The study aims to evaluate the contribution of a multi-targeted microbiotherapy at 12 weeks in depressed-patients in a situation of failure of a 1st line of antidepressant treatment and treated in add-on with a 2nd antidepressant, venlafaxine.

DETAILED DESCRIPTION:
Depression is the most common psychiatric illness and has major personal, societal and economic consequences.

Increase in the disease prevalence is significantly associated with certain somatic pathologies, including metabolic diseases and functional intestinal disorders. From a therapeutic point of view, approximately 2/3 patients are not in remission after first-line antidepressant treatment. Moreover, 20 to 30% patients resist at all the therapeutic strategies classically proposed in this indication.

The identification of new therapeutic strategies is therefore a major challenge, especially for patients with chronic depression resistant to standard treatments.

Various research studies have shown the involvement of inflammatory mechanisms in depression. Thus, the increase in the disease prevalence is significantly associated with certain somatic pathologies, in particular metabolic diseases, a certain number of which are linked to abnormalities of the intestinal microbiota. In this context, the use of probiotics is interesting because some have antidepressant effects, anti-inflammatory and metabolic properties. However, even if a few studies have shown an antidepressant effect of probiotics with improvement of biological markers of inflammation, it seems that the use of probiotics alone is not sufficient for lasting results on depressive symptoms.

The PROMOOD clinical research project fits into this context. We propose to carry out a multicenter clinical study with the product developed by GYNOV (GynMDD® multitarget compound with 3 active ingredients: an amino acid (L-glutamine), an ingredient purified from a plant extract (Cavacurmine) and a probiotic (Lactobacillus rhamnosus GG). In a preclinical study carried out at the CNRS on 144 mice, a synergy of action between these 3 ingredients was demonstrated on the anxio-depressive systems, resulting in an improvement far greater than the expected effect of composition and comparable to a reference injectable antidepressant (clomipramine).

In theses context, the microbiotherapy proposed in this project is very original because:

* a multi-target approach targeting several mechanisms of action: intestinal permeability, glutamine/glutamate/GABA cycle, insulin resistance, immunomodulation, oxidative stress;
* prospect of an optimization/simplification of care;
* It is very acceptable for patients both from the point of view of tolerance and from the economic point of view.

With a phase II, prospective, multicenter design, this study aims to evaluate the contribution and the tolerance of a multi-targeted microbiotherapy in addition to venlafaxine, in a second-line antidepressant treatment. The treatment will be delivered during 12 weeks.

Baseline measures will be compared to those obtained during the treatement administration (every week) and after the treatment administration (every week for the next 12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unipolar MDD (Diagnostic and Statistical Manual of Mental Disorders V [DSM-V], QIDS-C16≥15)
* No response at a first antidepressant
* under venlafaxine
* Signed informed consent form
* Subjects affiliated to or beneficiary from a French social security regime

Exclusion Criteria:

* Contraindications to probiotic administration
* Allergy to one of the compounds of the multi-target probiotic or the placebo
* consuming probiotic-based dietary supplements
* Patient with other psychiatric disorders, except social anxiety disorder, generalized anxiety disorder and nicotine use disorder
* Patient with a serious and/or progressive medical condition, including chronic inflammatory pathologies or autoimmune diseases requiring long-term anti-inflammatory treatment (including corticosteroid therapy) or immunosuppressant.
* Patient with a recent infectious episode likely to require antibiotic therapy.
* Patient presenting with a suicidal risk assessed by the suicide item of the QIDS-C16 scale (score item 12 of the QIDS-C16 >2)
* Other concomitant antidepressant and/or lithium and/or anti-inflammatory treatment for the duration of the study
* Subject under measure of protection or guardianship of justice
* Subject beneficiary from a legal protection regime
* Subject unlikely to cooperate or low cooperation stated by investigator
* Subject not covered by social security
* Pregnant woman
* Subject being in the exclusion period of another study or provided for by the "National Volunteer File

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Quick Inventory of Depressive Symptomatology (QIDS-C16) at 12 weeks | baseline (Day 0), Week 12 (W12) post-treatment
  The QIDS-C16 is a 16-item scale that is clinician-rated; it is designed to assess the severity of depressive symptoms. The QIDS-C16 total score ranges from 0-27. Scores ranging from 0 to 10 correspond with no to mild depression, while scores >/= 11 correspond to moderate to severe depression. A negative change indicates improvement in the subject's depression, and a positive change indicates a worsening of the subject's depression.

SECONDARY OUTCOMES:
Change from Severity of depressive symptoms evaluated by the clinician | baseline (Day 0), at the end of therapy (week 12 (W12)
  The QIDS-C16 was derived from specified items in the IDS-C30, clinician-rated scale to assess the severity of a participant's depressive symptoms. Total scores range from 0-27, with a score of 0 indicating no depression and a score of 27 indicating the most severe depression. Negative change from baseline values indicate improvement in the severity of depression.
Change from Severity of depressive symptoms evaluated by the patient | baseline (Day 0), at the end of therapy (week 12 (W12)
  Score achieved on the validated self-reported (QIDS-SR16) evaluating the severity of depressive symptoms. QIDS-SR-16 is a standard questionnaire "The Quick Inventory of Depressive Symptomatology" (16-Item) (Self-Report). This covers questions on falling asleep, sleep during the night, waking up , sleeping too much, feeling sad ,appetite, weight, concentration , how they view themselves, thoughts of death and suicide, general interests, energy levels, feeling slowed down , feeling restless.
Evaluation of treatment observance | baseline (Day 0), at the end of therapy (week 12 (W12)
  A treament observance book was complied by patient during the 12 weeks of therapy
Change from Health related Quality of Life (HrQoL) | baseline (Day 0), at the end of therapy (week 12 (W12)
  HrQOL will be assessed using health status measures of the EuroQuality of Life Five Dimensions (EQ-5D-5L)
Change from anxiety | baseline (Day 0), at the end ot therapy (week 12 (W12)
  anxiety assessed using Brief Anxiety Scale of Tyrer (BAS)
Change from digestive health | baseline (Day 0), at the end ot therapy (week 12 (W12)
  digestive evaluation assessed by digestive health scale, scale developped by gastroenterlogists (https://www.worldgastroenterology.org/search?cx=005474681532606414716%3AWMX-367025812&cof=FORID%3A9&ie=UTF-8&q=digestive+health+evaluation)
Change from serum Inflammatory biological markers | baseline (Day 0), at the end ot therapy (week 12 (W12)
  inflammatory inflammatory levels (CRP, Il-1b, Il-6 and TNF-a) in blood samples
Change from Biological markers of intestinal dysbiosis | baseline (Day 0), at the end ot therapy (week 12 (W12)
  zonulin and serobank levels in blood samples
Change from Metagenomic shotgun sequencing of gut microbiota | baseline (Day 0), at the end ot therapy (week 12 (W12)
  preforming metagenomic shotgun sequencing of fecal DNA to determine the changes in the intestinal microbiota composition, diversity and functionality

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel HAFFEN, MD PhD, Principal Investigator — CHU de Besançon
Locations (4):
- France (4):
  - Emmanuel HAFFEN, Besançon
  - Centre Hospitalier Spécialisé Charles Perrens, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor / APHP, Créteil

IPD SHARING:
Plan to Share IPD: No